CLINICAL TRIAL: NCT01396109
Title: A Prospective, Multicenter Trial to Compare GYNECARE PROSIMA* Pelvic Floor Repair System Procedure With Modified Total Pelvic Floor Reconstruction Surgery Concomitantly With TVH to Treat Symptomatic POP-Q Stage III Uterine Prolapse
Brief Title: GYNECARE PROSIMA* Procedure Versus Modified Total Pelvic Floor Reconstructive Surgery for Uterine Prolapse Stage III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pumch-gyn-01
Record Dates: First submitted 2011-07-13; First posted 2011-07-18 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2011-03

CONDITIONS: Uterine Prolapse; Stage III
MeSH Terms: conditions — Uterine Prolapse | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Active Comparator): Intervention: Procedure: TVH and GYNECARE PROSIMA* Pelvic Floor Repair System
  Interventions: Procedure: Procedure: TVH and GYNECARE PROSIMA* Pelvic Floor Repair System
- Group II (Active Comparator): Intervention: Procedure: TVH and Modified Pelvic Floor Reconstruction Surgery with Mesh
  Interventions: Procedure: Procedure: TVH and Modified Pelvic Floor Reconstruction Surgery with mesh

INTERVENTIONS:
Procedure: Procedure: TVH and GYNECARE PROSIMA* Pelvic Floor Repair System — Subjects of this group were submitted to surgical treatment with GYNECARE PROSIMA* Pelvic Floor Repair System concurrently with transvaginal hysterectomy.
  Arms: Group I
Procedure: Procedure: TVH and Modified Pelvic Floor Reconstruction Surgery with mesh — Subjects of this group were submitted to surgical treatment of Modified Pelvic Floor Reconstruction Surgery with mesh concurrently with transvaginal hysterectomy.
  Arms: Group II

SUMMARY:
Pelvic Organ prolapse (a feeling of bulge in the vagina) may cause some distressing symptoms such as loss of control of the bowel or bladder, and may also cause problems with patient's sex life. The primary treatment is surgery, sometimes a mesh is placed in the pelvis to support the weakened tissues, but mesh implants can cause complications.

This study is designed to determine the effectiveness and safety of GYNECARE PROSIMA* pelvic floor repair system compared with the modified total pelvic floor reconstructive surgery with mesh for the treatment of uterine prolapse.

Patients enrolled into the study will be followed up for up to 3 years after surgery. Evaluation will take place during surgery and postoperative visit. Stage of prolapse before and after surgery, patient satisfaction through quality of life and sexual function questionnaires before and after surgery, and peri-operative complication rates will be evaluated.

DETAILED DESCRIPTION:
Pelvic organ prolapse is a common problem. The high rate of failure has led to an increasing use of synthetic grafts to augment vaginal repair procedures to obtain more durable results. In 2005, the investigators began to perform modified pelvic floor reconstruction surgery with mesh. The nation-wide multicenter prospective clinical trial data showed that it was safe, efficient and cost-effective. No severe intraoperative complications were recorded and the recurrence rate after 1 year follow-up was 8.1%. Quality of life improved significantly from the baseline, while the sexual function did not change.

The GYNECARE PROSIMA* system is a new technique. It provides a simplified unanchored mesh repair, avoiding the need for dissection outside the pelvic cavity and avoids passage of suture and instruments through the obturator foramen and sacrospinous ligament, thus making surgery much simpler to perform and reduces the risk of the specific complications that can occur with suture placement or tunneling. 1-year anatomic and functional outcomes of international multicenter prospective study for POP-Q Stage I I-III pelvic organ prolapse showed the objective success rate was 76.9%, pelvic symptoms, quality of life, and sexual function improved significantly from baseline.

In clinical practice, many women have symptomatic POP-Q Stage III uterine prolapse, which requires surgical correction. They are relatively young, and therefore care more about the long-term outcomes and quality of life after procedure. The purpose of this multicenter, prospective, and comparative study is to evaluate the effectiveness and safety of these two procedures concomitantly performed with vaginal hysterectomy (TVH) in the treatment of symptomatic POP-Q Stage III uterine prolapse in China.

ELIGIBILITY:
Inclusion Criteria:

* Candidates with symptomatic uterine prolapse of ICS POP-Q Stage III(with any degree of vaginal prolapse), suitable for surgical repair.
* Vaginal hysterectomy will be performed concurrently.
* Without stress urinary incontinence or occult stress urinary incontinence with no need of mid-urethral sling procedures for incontinence to be performed.
* Age ≥ 60 years.
* Agrees to participate in the study, including completion of all study-related procedures, evaluations and questionnaires, and documents this agreement by signing the Ethics Committee / IRB approved informed consent.

Exclusion Criteria:

* Additional surgical intervention concurrent to the procedure (e.g. sacrocolpopexy, paravaginal repair, tubal sterilisation).
* Previous repair of pelvic organ prolapse involving insertion of mesh.
* Experimental drug or experimental medical device within 3 months prior to the planned procedure.
* Active genital, urinary or systemic infection at the time of the surgical procedure. Surgery may be delayed in such subjects until the infection is cleared.
* Coagulation disorder or on therapeutic anticoagulant therapy at the time of surgery.
* History of chemotherapy or pelvic radiation therapy.
* Systemic disease known to affect bladder or bowel function (e.g. Parkinson's disease, multiple sclerosis, spinal cord injury or trauma).
* Current evaluation or treatment for chronic pelvic pain (e.g. interstitial cystitis, endometriosis, coccydynia, vulvodynia).
* Nursing or pregnant or intends future pregnancy.
* Chronic cough not well-controlled.
* BMI≥30.
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Anatomical improvement according to POP-Q score. | 4 weeks
Anatomical improvement according to POP-Q score. | 6 months
Anatomical improvement according to POP-Q score. | 12 months
Anatomical improvement according to POP-Q score. | 2 years
Anatomical improvement according to POP-Q score. | 3 years

SECONDARY OUTCOMES:
Hospital data including operative time, estimated blood loss, length of stay, maximum temperature, time of voiding recovery. | At discharge, an expected average of 5 days after operation.
Pain score measured using Visual Analog Scale (VAS). | 24 hours post surgery and at the 3-4 week visit
Presence/absence of complications (composite score). | Up to 6 weeks.
  The occurrence (in the per-operative phase or within 6 weeks post-op) of at least one of the following: 1) bleeding complications; 2) infectious complications; 3) any wound caused by a surgeon movement: bladder, ureteral, or vascular injuries; 4)medical complications: deep vein thrombosis, pulmonary embolism and etc.Complications will be categorized using the Dindo surgical complication grading scale.
Change from baseline in PFIQ-7 scores. | 6 months, 12 months, 2 years and 3 years.
In subjects sexually active at baseline, assessment of sexual function using PISQ-12 (mean scores and change from baseline) | 6 months, 12 months, 2 years and 3 years.
Subject global impression assessed on a 5 point Likert scale | 6 months, 12 months, 2 years and 3 years.
Presence/absence of complications (composite score) | Up to 3 years.
  Long-term negative outcomes of the surgical procedure will also be recorded until 3 years after surgery. For example, mesh erosion, de novo urinary incontinence, de novo dyspareunia and overall failure rate. Complications will be categorized using the Dindo surgical complication grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (10):
- China (10):
  - Hefei Maternity and Child Health Hospital, Hefei, Anhui
  - Gansu Maternity and Child Health Hospital, Lanzhou, Gansu
  - Hebei Provincial Hospital, Shijiazhuang, Hebei
  - the First Affliliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuxi Maternal and Child Health Hospital, Nanjing Medical University, Wuxi, Jiangsu
  - Maternal and Child Health Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Laizhou Municipal People's Hospital, Laizhou, Shandong
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing